CLINICAL TRIAL: NCT00505843
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Period Crossover Study to Evaluate Effectiveness of Single-Dose MK0657 in Combination With Levodopa on Motor Symptoms and Dyskinesias in Patients With Parkinson's Disease
Brief Title: A Study of MK0657 in Parkinson's Disease Patients (0657-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0657-006; MK0657-006; 2007_524
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 4-methylbenzyl 3-fluoro-4-((pyrimidin-2-ylamino)methyl)piperidine-1-carboxylate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): 7mg MK0657 capsules + >/=1.0 mg/kg/hr dose of levodopa.
  Interventions: Drug: MK0657; Drug: Comparator: levodopa; Drug: Comparator: carbidopa
- 2 (Other): 7mg MK0657 Pbo capsules + >/=1.0 mg/kg/hr dose of levodopa.
  Interventions: Drug: Comparator: Placebo (unspecified); Drug: Comparator: levodopa; Drug: Comparator: carbidopa

INTERVENTIONS:
Drug: MK0657 — 7mg MK0657 capsules
  Arms: 1
Drug: Comparator: Placebo (unspecified) — 7mg MK0657 Pbo capsules
  Arms: 2
Drug: Comparator: levodopa — levodopa >/=1.0 mg/kg/hr dose of levodopa. levodopa infusions will occur over a 2 hour period
Drug: Comparator: carbidopa — carbidopa 25mg administered 3 times: at 1 hour before levodopa infusion and at 1 and 3 hours after the start of levodopa infusion.

SUMMARY:
In this clinical trial, the safety of MK0657 when given with levodopa will be assessed in patients with Parkinson's Disease. This study will also measure the effectiveness of MK0657, when given in combination with levodopa, to improve motor symptoms and ameliorate dyskinesias (uncontrolled movements of a part of the body) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease patients between the ages of 40 and 80 inclusive
* Patient is in general good health based on screening assessments
* Patient is willing to discontinue anti-parkinson's medications at least 8 hours prior to dosing
* Patient is levodopa responsive with levodopa-induced peak-dose dyskinesias
* Patient taking selective serotonin inhibitors (SSRIs), sleep medications and neuroleptics, have been on a stable dose for at least 30 days and has not experienced any CNS-related side effects
* Patient is not a heavy smoker or drinker

Exclusion Criteria:

* Patient has atypical Parkinson's syndrome due to drugs, identified metabolic and/or neurologic disorders, encephalitis, or other degenerative syndrome
* Patient has known intolerance or hypersensitivity to levodopa or carbidopa
* Patient has been on anticholinergics or memantine within 30 days prior to dosing
* Patients have a history of the following: seizure disorder, stroke or head trauma, pronounced cognitive impairment, psychiatric disorder, cardiovascular disease, cancer, diabetes as defined by HbA1c of greater than 8%
* Patient has a systolic BP or less than 80 mm Hg or greater than 150 mm Hg

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed for up to 8 hours by the Unified Parkinson's Disease Rating Scale-Motor Examination and a modified AIMS dyskinesia scale | 45 Days

SECONDARY OUTCOMES:
Safety and Tolerability | 45 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Addy C, Assaid C, Hreniuk D, Stroh M, Xu Y, Herring WJ, Ellenbogen A, Jinnah HA, Kirby L, Leibowitz MT, Stewart RM, Tarsy D, Tetrud J, Stoch SA, Gottesdiener K, Wagner J. Single-dose administration of MK-0657, an NR2B-selective NMDA antagonist, does not result in clinically meaningful improvement in motor function in patients with moderate Parkinson's disease. J Clin Pharmacol. 2009 Jul;49(7):856-64. doi: 10.1177/0091270009336735. Epub 2009 Jun 2. PMID 19491335
- [Derived] Herring WJ, Assaid C, Budd K, Vargo R, Mazenko RS, Lines C, Ellenbogen A, Verhagen Metman L. A Phase Ib Randomized Controlled Study to Evaluate the Effectiveness of a Single-Dose of the NR2B Selective N-Methyl-D-Aspartate Antagonist MK-0657 on Levodopa-Induced Dyskinesias and Motor Symptoms in Patients With Parkinson Disease. Clin Neuropharmacol. 2017 Nov/Dec;40(6):255-260. doi: 10.1097/WNF.0000000000000241. PMID 29059133